CLINICAL TRIAL: NCT03133533
Title: Laparoscopic Versus Robot-assisted Inguinal Hernia Repair: The Immediate, Intermediate, and Long Term Outcome Differences. A Single Institution Randomized Controlled Trial
Brief Title: Laparoscopic Versus Robot-assisted Inguinal Hernia Repair: A Single Institution Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI on an extended leave of absence.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601494
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Hernia, Inguinal
Keywords: robot-assisted
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either laparoscopic or robot-assisted repair of inguinal hernia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic (Active Comparator): laparoscopic inguinal hernia repair
  Interventions: Procedure: laparoscopic repair
- robot-assisted (Active Comparator): robot-assisted inguinal hernia repair
  Interventions: Procedure: robot-assisted repair

INTERVENTIONS:
Procedure: laparoscopic repair — Surgical inguinal hernia repair using laparoscopic approach.
  Arms: laparoscopic
Procedure: robot-assisted repair — Surgical inguinal hernia repair using robot-assisted approach.
  Arms: robot-assisted

SUMMARY:
Randomized trial to compare outcomes of laparoscopic and robot assisted inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia repair is a very common surgical operation. Both laparoscopic and robot-assisted operations are considered acceptable. However, there is no clear indication for a particular approach. No prospective trial has been conducted so far to establish superiority of one approach over the other. The Investigator believes each approach has unique characteristics and may offer advantages over the other in the right population group. The Investigator will randomly assign patients in two arms according to the surgical approach, whether laparoscopic or robot-assisted. The Investigator will collect preoperative characteristics, intraoperative variables, and postoperative outcomes. The Investigator will compare all variables to establish differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* surgeon determined need for inguinal hernia repair

Exclusion Criteria:

* < 18 years of age
* > 99 years of age
* medical indication for open repair

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Operative time | Immediate perioperative time
  Time from start to finish of procedure, procedure start and stop times as recorded by anesthesia.

SECONDARY OUTCOMES:
Postoperative pain score | Until 5 year postoperative
  Abdominal pain at rest and on moving (recumbent to the upright position), will be assessed using 0-10 Numeric Pain Rating Scale preoperatively (baseline), and at 24 hours, 30 days, one and five years postoperatively.

OTHER OUTCOMES:
Complications | From immediately post-operative until year five following surgical inguinal hernia repair.
  Postoperative 30 day complication rates will be recorded prospectively. All complications (including multiple occurrences per patient) will be recorded and graded per the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Latzko, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No